CLINICAL TRIAL: NCT06006078
Title: Does Use of a Facemask Reduce the Risk of Aerosolization During Anesthesia Assisted Upper Endoscopic Procedures: A Randomized Controlled Trial
Brief Title: Aerosolization During Upper Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Lembo (Other)
Responsible Party: Sponsor-Investigator, Anthony Lembo, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-641
Record Dates: First submitted 2023-05-16; First posted 2023-08-23 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Infectious; Gastro-Intestinal Disorder; Safety Issues
MeSH Terms: conditions — Communicable Diseases; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: One group of patients will be randomly assigned to receive an endoscopic facemask and one group of patients will undergo endoscopy without a facemask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Endoscopic Facemask (Active Comparator): Patients undergoing endoscopy with the use of an endoscopic facemask
  Interventions: Device: Endoscopic Patient Facemask
- No Endoscopic Facemask (No Intervention): Patients undergoing endoscopy without an endoscopic facemask

INTERVENTIONS:
Device: Endoscopic Patient Facemask — A commonly used endoscopic patient facemask that is normally used for oxygen delivery during endoscopy will be tested in this trial as a potential intervention for decreasing particle aerosolization
  Other Names: POM Mask
  Arms: Endoscopic Facemask

SUMMARY:
Given the current Covid-19 pandemic alongside the lack of evidence on aerosolization during upper endoscopy the investigators are conducting a randomized controlled trial seeking to assess both the level of aerosolization that occurs during these procedures along with determining if utilization of an endoscopic patient face-masks reduces the level of aerosolized particles. The protocol includes the use of a commercially available particle counter the investigators are employing for the measurement of aerosols before, during, and after anesthesia assisted upper endoscopic procedures. The investigators are recruiting patients undergoing these procedures with a target of 30 patients undergoing endoscopy without a facemask and 30 patients undergoing endoscopy with one.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective upper endoscopic procedures (upper endoscopy, ERCP, endoscopic ultrasound) with monitored anesthesia care at main campus Cleveland Clinic inpatient endoscopy unit.

Exclusion Criteria:

* Any patient requiring endotracheal intubation
* Pregnant patients
* Emergency procedures
* Patients who require use of a facemask before or during the procedure due to medical necessity
* Patients under the age of 18
* Non-English speaking individuals
* Patients unable to provide consent.
* Any procedure done outside the designated procedure room.
* If in the opinion of the anesthesiologist, a subject who was randomized to the control arm requires placement of the procedural mask to augment oxygenation, the subject will be removed from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Vargo, MD, Principal Investigator — Physician
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endoscopic Facemask | No Endoscopic Facemask
Started | 27 | 30
Completed | 27 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endoscopic Facemask | No Endoscopic Facemask | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (17.0) | 59.6 (16.7) | 59 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 33
  Male | 15 | 9 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Aerosolization of Particles During Upper Endoscopy
Description: Comparing the aerosolization of particles of six different sizes [0.3μm, 0.5μm, 1μm, 2μm, 5μm and 10μm] during endoscopy between patients using an endoscopic facemask to those without.
Time Frame: Start of endoscopy through the end of endoscopy
Population: The data will be analyzed via stratification by particle size as a as a volumetric measurement of density: the number of particles per unit volume.
Measure: Least Squares Mean (95% Confidence Interval); unit: particle count per cubic ft
Arm/Group | Endoscopic Facemask | No Endoscopic Facemask
Number analyzed (Participants) | 27 | 30
particle count per cubic ft
  less than 0.3 μm | 9.86 [9.62 to 10.1] | 9.87 [9.65 to 10.1]
  0.3- 0.5 μm | 6.93 [6.66 to 7.21] | 7.05 [6.8 to 7.31]
  0.5- 0.7 μm | 5.63 [5.32 to 5.93] | 5.49 [5.19 to 5.78]
  0.7- 1.0 μm | 6.33 [6.1 to 6.57] | 6.34 [6.12 to 6.56]
  1.0- 5.0 μm | 4.73 [4.62 to 4.84] | 4.74 [4.63 to 4.84]
  5.0 - 10 μm | 4.78 [4.68 to 4.88] | 4.71 [4.61 to 4.8]

ADVERSE EVENTS:
Description: Adverse events were not collected for the study.
Arm/Group | Endoscopic Facemask | No Endoscopic Facemask
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT06006078/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT06006078/ICF_001.pdf